CLINICAL TRIAL: NCT01218139
Title: Analysis of Peripheral Nerve Sheath Tumors in Neurofibromatosis Type 1 Patients
Brief Title: Analysis of Peripheral Nerve Sheath Tumors (PNSTs) in Neurofibromatosis Type 1 (NF1) Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Eric Legius, KUL
Other Study IDs: LEGIUS_001
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-10

CONDITIONS: Neurofibromatosis Type 1
Keywords: neurofibroma; MPNST; array CGH; sequencing
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma; Neurofibrosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Neurofibromatosis type 1 (NF1) is a frequent, autosomal dominant disorder caused by heterozygous mutations (intragenic or microdeletion) of the NF1 tumor suppressor gene (chr.17q11.2). One of the clinical features is the development of benign and malignant tumors. The most common benign tumors in these patients are tumors of the peripheral nerve sheath, named neurofibromas (cutaneous, subcutaneous and plexiform). Every NF1 patient has a life time risk of 8 to 13% of developing a malignant peripheral nerve sheath tumor (MPNST) out of a pre-existing neurofibroma. In patients with a NF1 microdeletion (5% of NF1 patients), this risk is even twice as high compared to patients with an intragenic mutation. MPNSTs lead to a bad prognosis for the patient, with an overall five-year survival of less than 25%. To know more about the development and progression of these tumors, they will be screened by microarray comparative genome hybridization (Leuven) and full exome sequencing (Leuven). Further experiments will be done in cooperation (bidirectional) with the foreign labs of Victor Mautner (Germany), André Bernards (USA), Karen Cichowski (USA) and Yuan Zhu (USA).

For all these experiments, we will make use of tumoral rest material removed from NF1 patients.

DETAILED DESCRIPTION:
Introduction Neurofibromatosis type 1 (NF1) is an autosomal dominant disorder occuring in 1 out of 3500 living newborns. The disease is caused by heterozygous mutations of the NF1 gene, located on chromosome 17q11.2. The NF1 gene encodes the tumor suppressor neurofibromin, a negative regulator of the RAS/MAPK pathway. In approximately 95% of patients, the heterozygous mutation is intragenic. The remaining 5% of patients are carrier of a microdeletion, mostly the type 1 deletion, in which apart from the NF1 gene, 14 additional protein coding genes are located.

Clinically, NF1 patients have café-au-lait maculae, freckling, Lisch nodules and neurofibromas. Also cognitive problems, bone lesions and optic pathway gliomas are common in these patients.

Neurofibromas are benign neoplasms of the peripheral nerve sheath, which appear everywhere on the body of almost every NF1 patient. Neurofibromas are composed of different cell types like Schwann cells, fibroblasts, mast cells and perineurial cells. If in Schwann cells of NF1 patients the wild-type NF1 allele is inactivated in a heterozygous microenvironment, a neurofibroma will be formed. There are 3 types of neurofibromas: cutaneous, subcutaneous and plexiform. Cutaneous and subcutaneous neurofibromas appear during adolescence as isolated nodules in or under the skin, respectively. Plexiform neurofibromas are congenital and can spread along a large segment of a peripheral nerve. NF1 microdeletion patients have in general more neurofibromas and they appear at a younger age.

Every NF1 patient has a life time risk of 8 to 13% to develop a malignant peripheral nerve sheath tumor (MPNST) out of a pre-existing (plexiform) neurofibroma. This risk is even twice as high for NF1 microdeletion patients compared to patients with an intragenic mutation. MPNSTs are difficult to diagnose in early phase because of the large number of tumors and diverse locations. These tumors infiltrate easily in surrounding tissue and frequently give rise to metastases. At this moment, the only available treatment is surgical removal of these MPNSTs. Complete resection is often difficult due to the size of the tumors and the location on important nerves. The five-year survival of patients with MPNSTs is less than 25%.

Research protocol All NF1 patients are linked to the UZ Leuven. Their follow-up is done by Prof. Dr. Eric Legius. When the patient is suspected of having a MPNST, the patient is referred to the surgeon of the clinical oncology department, respectively. Also neurofibromas are removed when they are causing problems for the patient. As part of the different tumor care programs in our hospital, a tumor piece is sent from pathology to the centre for human genetics for routine genetical analysis, like karyotyping. In the lab for neurofibromatosis research, the rest material is frozen as tumor pieces and as dissociated cells for research purposes. The samples are stored in a database system that is accessible only for the neurofibromatosis research group. In cooperation with the group of Victor Mautner and Karen Cichowski, the tumor database was further completed with NF1 tumor material and cell lines. The latter samples were coded and could be used as part of our collaboration.

Experimental approach In literature, little is known about the development of a MPNST out of a neurofibroma. In this study we want to gain insight into this process, which can in the end lead to a better diagnosis and treatment of NF1 patients with MPNSTs. For this purpose, only the frozen rest material of neurofibromas and MPNSTs will be used.

At first, DNA will be extracted from the frozen tumor pieces (neurofibromas and MPNSTs). Together with blood DNA (also rest material), the tumor DNA will be screened with microarray genomic hybridization. This technique allows us to check for chromosomal abnormalities, like amplifications and deletions, with a much higher resolution than traditional cytogenetics. In that way, we can look for recurrent alterations within a certain tumor type and for similarities and differences between benign and malignant tumors.

Secondly, the group of MPNSTs will be subdivided in tumors derived from NF1 microdeletion patients and tumors from patients with an intragenic mutation. Recurrent chromosomal gains and losses will be compared between the 2 groups. This will show us if the mechanism of tumor development and progression is different in NF1 microdeletion patients. In cooperation with the group of André Bernards and Karen Cichowski, we will try to elucidate the role of the NF1 microdeletion in the development of neurofibromas. Our group will collect all tumor samples and grow Schwann cells and fibroblasts out of these tumors. The frozen vials with tumor pieces and cultured cells will be encoded and provided to these labs as part of our collaboration.

Subsequently, the DNA derived from 10 different tumors (neurofibromas and MPNSTs) and matching blood DNA will be analyzed by 'full exome sequencing' to check for mutations in all coding exons.

In collaboration with the group of Yuan Zhu, tumor samples will be sent and retrieved in an encoded way.

This study is performed by Eline Beert, PhD student in the lab for neurofibromatosis research, as part of achieving the degree of 'Doctor in Biomedical Sciences', with Prof. Dr. Eric Legius as promotor and main researcher. Only the Catholic University of Leuven and other foreign universities, but no commercial partners (like companies) will participate in this study. The results obtained from the described experiments have to be considered as pure scientific information and none will be reported to the patients.

ELIGIBILITY:
Inclusion Criteria:

NF1 patient

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: population of NF1 patients, seen by prof. Eric Legius, who are having surgery to remove a tumor
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Legius, MD PhD, Principal Investigator — KU Leuven
Locations (1):
- KUL, Leuven, Vlaams-Brabant, Belgium